CLINICAL TRIAL: NCT02455154
Title: Traditional Chinese Medicine as Preventive Method for Osteoporosis in Early Breast Cancer Patients Receiving Adjuvant Endocrine Therapy
Brief Title: Traditional Chinese Medicine as Preventive Method for Osteoporosis Induced by Adjuvant Endocrine Therapy
Acronym: COAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Kunwei Shen, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RJBC1502
Record Dates: First submitted 2015-05-14; First posted 2015-05-27 (Estimated); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer; Osteoporosis
Keywords: Chinese Traditional Medicine; Osteoporosis; adjuvant endocrine therapy; early breast cancer
MeSH Terms: conditions — Breast Neoplasms; Osteoporosis | interventions — Letrozole; xian ling gu bao

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Letrozole (Placebo Comparator): Early Breast Cancer patients receiving adjuvant endocrine therapy
  Adjuvant Endocrine Therapy: letrozole 2.5 mg qd po.
  Interventions: Drug: Letrozole
- Letrozole + Xinglinggubao (Active Comparator): Early Breast Cancer patients receiving adjuvant endocrine therapy plus Xianlinggubao
  Adjuvant Endocrine Therapy: letrozole 2.5 mg qd po.
  Xinglinggubao: 0.5g bid po
  Interventions: Drug: Letrozole; Drug: Xianlinggubao
- Letrozole + Zhongyaofufang (Active Comparator): Early Breast Cancer patients receiving adjuvant endocrine therapyplus Zhongyaofufang (Traditional Chinses Medicine)
  Adjuvant Endocrine Therapy: letrozole 2.5 mg qd po.
  Zhongyaofufang: qow po
  Interventions: Drug: Letrozole; Drug: Zhongyaofufang

INTERVENTIONS:
Drug: Letrozole — Letrozole endocrine therapy for 2.5mg qd po.
  Other Names: L
Drug: Zhongyaofufang — Traditional Chinese Medicine for patients with Osteoporosis
  Other Names: Z
  Arms: Letrozole + Zhongyaofufang
Drug: Xianlinggubao — Traditional Chinese Medicine for patients with Osteoporosis
  Other Names: X
  Arms: Letrozole + Xinglinggubao

SUMMARY:
To test the efficacy of two Traditional Chinese Medicine in preventing osteoporosis in patients receiving adjuvant endocrine therapy.

DETAILED DESCRIPTION:
Breast cancer is the most common malignant tumor in female wolrdwide. Results from clinical trials like ATAC trial have demonstrated the efficacy of AIs in postmenopausal breast cancer patients. Meanwhile it may cause a certain rate of osteoporosis in postmenopausal patients. The aim of this trial is to test the efficacy of two traditional Chinese medicine in preventing osteoporosis in patients receiving adjuvant endocrine therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive breast cancer;
* Post-surgery, primary lesion been removed;
* Post-Menopausal patients or pre-menopausal patients who will receive ovarian function suppression;
* Histologically confirmed ER and/or PR positive ;
* Receiving adjuvant AIs therapy in the following one years;
* Leukocyte ≥ 3*10(9)/L; Platelets ≥ 75*10(9)/L;
* Serum glutamate oxaloacetate(AST/SGOT) or serum glutamic-pyruvic transaminase(ALT/SGPT) <2.5 times of upper limit of normal range;
* Serum creatinine/blood urea nitrogen(BUN) ≤ upper limit of normal (UNL) range;
* Written informed consent according to the local ethics committee equirements;

Exclusion Criteria:

* Metastatic Breast Cancer;
* Received Neo-Adjuvant Endocrine Therapy;
* History of pelvic fracture or bone metabolic disease;
* Received drugs interfering bone metabolism in the last 12 months;
* Baseline Bone Mineral Density: T < -2SD;
* With other primary malignant disease;
* With severe non-malignant co-morbidity that will influence long-term follow up;
* Known severe hypersensitivity to any drugs in this study;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2015-05; Primary Completion 2019-02 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Change of Bone Mineral Density | 1 year
  The change of bone mineral density of the L2-L4 region of the spine and hip between pre- and post-endocrine therapy for one year

SECONDARY OUTCOMES:
Bone Frature Rate | 1 year
  the rate of bone fracture in patient receiving endocrine therapy
Bone Metabolism | 1 year
  The change of bone metabolism assessed by the scale of serum bone alkaline phosphatase, serum C-telopeptide and urineN-telopeptide between pre- and post-endocrine therapy for one year
Disease Free Survival | 1 year
  the rate of patients without disease

CONTACTS AND LOCATIONS:
Overall Officials: Kunwei Shen, MD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China